CLINICAL TRIAL: NCT04528030
Title: WAVE Trial in Premature Infants With Apnea of Prematurity Using a Simple, Non-invasive Vibratory Device to Study the Effectiveness in Supporting Breathing and General Stability
Brief Title: A UK Interventional Trial in Premature Infants With Apnea of Prematurity Using a Simple, Non-invasive Vibratory Device to Study the Effectiveness in Supporting Breathing and General Stability
Acronym: WAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inspiration Healthcare (Other)
Collaborators: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CRR-WAVE-122-CIP
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Apnea of Newborn; Hypoxia Neonatal; Bradycardia Neonatal
Keywords: cardio-respiratory stability; neonate; premature infant; proprioceptive stimulation; Apnoea of Prematurity; Medical Device
MeSH Terms: conditions — Asphyxia Neonatorum; Premature Birth; Apnea

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
  In the same subject there were 2 periods:
  OFF cycles (6 hours x 2): 'No intervention' period (no vibrations) - two 6 hour epochs - total of 12 hours of 'No intervention' ON cycles (6hours x 2). Experimental period (with vibrations) - two 6 hour epochs - total of 12 hours of 'vibration intervention'
  In the same subjects cardio-respiratory parameters will be continuously monitored through the 24 hour treatment period of 4 cycles- heart rate, respiratory rate and oxygen saturation were compared during the experimental period (vibration) and during the no intervention period (no vibration).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator analyzing the 4 cycles will not know whether it's an ON of OFF cycle during the 24 hour treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment starting with an on ON cycle (Other): The treatment will start ON cycle for 6 hours, followed by OFF cycle for 6 hours, followed by OFF cycle for 6 hours and finished with ON cycle for 6 hours.
  Interventions: Device: WAVE device
- Treatment starting with an on OFF cycle (Other): The treatment will start OFF cycle for 6 hours, followed by ON cycle for 6 hours, followed by OFF cycle for 6 hours and finished with ON cycle for 6 hours.
  Interventions: Device: WAVE device

INTERVENTIONS:
Device: WAVE device — WAVE applies a transcutaneous vibration to the soles of the foot and palms of the hand to elicit nerve signalling from pressure and other limb proprioceptor sensors to pontine, cerebellar, and medullary brain areas that coordinate limb movement and reflexively activate brain areas controlling breathing. The WAVE device is a battery-operated product to reduce the episodes of Apnoea of Prematurity by vibratory stimulation to the hand and foot.
  Other Names: limb proprioceptive stimulation; kinesthetic stimulation

SUMMARY:
Purpose of Study: Apnoea of Prematurity (AOP) is common, affecting the majority of infants born <34 weeks gestational age (GA). Apnea is accompanied by intermittent hypoxia (IH), which contributes to multiple pathologies, including retinopathy of prematurity (ROP), sympathetic ganglia injury, impaired pancreatic islet cell and bone development, and neurodevelopmental disabilities. Standard of care for AOP/IH includes prone positioning, positive pressure ventilation, and caffeine therapy. The objective of this device is to provide an adjunct to current AoP treatment to support breathing in premature infants by using a simple, non-invasive vibratory device placed over limb proprioceptor fibers, an intervention using the principle that limb movements facilitate breathing.

Methods Used: Premature infants (27+6 - 34+6 weeks GA) with clinical confirmed weeks with diagnosis of Apnoea of Prematurity. Caffeine therapy was not a reason for exclusion. Small vibration devices were placed on one hand and one foot and activated in a 6 hour ON/OFF sequence for a total of 24 hours. Heart rate, respiratory rate, oxygen saturation (SpO2), and breathing pauses were continuously collected.

DETAILED DESCRIPTION:
Aim: To study the effect of (WAVE Device) limb proprioceptive stimulation using a vibratory device on AoP events, intermittent hypoxic episodes (SpO2≤85%) and bradycardias(≤100bpm) in a premature infant with confirmed clinical diagnosis of apnea of prematurity (AoP).

The objective of the WAVE device is to provide an adjunct to current care to provide support in apnea of prematurity (AOP). Recurrent apnea and accompanying resultant intermittent hypoxic (IH) episodes are significant concerns commonly encountered in premature infants, and optimal management is a challenge to neonatologists. AoP is defined as >20s breathing pause OR breathing pause of 10-20sec with clinical signs of Bradycardia (≤100bpm) and/or desaturation (≤85% SpO2) in infants born less than 37 weeks of gestation. When these pauses are longer (> 20s), they are frequently prolonged by obstructed inspiratory efforts, most likely secondary to loss of upper airway tonic activity. In extremely low birth weight (ELBW) infants, the incidence of IH progressively increases over the first 4 weeks of postnatal life, followed by a plateau and subsequent decline between 6-8 weeks.

The incidence of AOP correlates inversely with gestational age and birth weight. Nearly all infants born <29 weeks gestation or <1,000 g, 54% at 30 to 31 weeks, 15% at 32 to 33 weeks, and 7% at 34 to 35 weeks gestation exhibit AOP (2). Both animal and human evidence show that immature or impaired respiratory control and the resultant IH exposure contribute to a variety of pathophysiologic issues via pro-inflammatory and/or pro-oxidant cascade as well as cellular mechanisms, e.g., apoptosis, leading to acute and chronic morbidities (e.g. retinopathy of prematurity, altered growth and cardiovascular regulation, disrupting zinc homeostasis which hampers insulin production and there by predisposing to diabetes in later life, cerebellar injuries and neurodevelopmental disabilities).

Current standard of care for AOP includes prone positioning, continuous positive airway pressure (CPAP) or nasal intermittent positive pressure ventilation (NIPPV) to prevent pharyngeal collapse and alveolar atelectasis, and methylxanthine therapy (caffeine, theophylline), which is the mainstay of treatment of central apnea. Apart from prone positioning, none of these interventions are optimal for early development. CPAP masks will distort the bony facial structure in early development, and methylxanthine interventions pose serious questions of neural development interactions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Gestational age > 27+6weeks, < 34+1 weeks
* Diagnosis of apnoea of prematurity (AOP) on clinical observations (atleast 4 AoP episodes and atleast one ABD event (equal and less 85% SpO2)- define clearly).
* Caffeine treatment will not be an exclusion. If babies are on caffeine they need on maintenance dose for atleats 48 hours. (72hours after first dose of caffeine (Infant must be on maintenance dose)
* During screening baby must demonstrate >4 AoP/1 ABD events
* Minimum 48 hours after extubation.

Exclusion Criteria:

* Inotropes
* Infants with major congenital anomalies/malformations which will influence central nervous system and long-term outcomes in these infants, such as cardiac anomalies (except for Patent Ductus Arteriosus or Ventricular Septal Defect) or major neurological malformations, like meningoencephalocele, holoprosencephaly
* Neonates who have apnoea from airway issues like laryngomalacia or tracheomalacia.
* Neonates with a history of hypoxic-ischemic encephalopathy or Grade IV intraventricular haemorrhage
* Infants that are currently intubated and invasive ventilation
* Congenital skin malformations, skin conditions due to recurrent illness (microcirculation concerns).
* Patients being treated for sepsis.

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Compare the cumulative burden of AoP with or without WAVE stimulation | 24 hours
  The primary objective is to compare the cumulative duration of breathing pauses related to Apnoea of Prematurity (AoP) between periods of presence and absence of tactile vibratory device stimulation as adjunct to standard care.

SECONDARY OUTCOMES:
Compare the number of AoP events. | 24 hours
  To compare the number of AoP events between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the number of desaturations (SpO2<86%) events | 24 hours
  To compare the number of desaturations (SpO2<86%) events between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the cumulative depth of desaturations. | 24 hours
  To compare the cumulative depth of desaturations (SpO2<86%) between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the cumulative duration of desaturations (SpO2<86%) events. | 24 hours
  To compare the cumulative duration of desaturations (SpO2<86%) between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the number of bradycardia events. | 24 hours
  To compare the number of bradycardia events between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the cumulative depth of bradycardia events. | 24 hours
  To compare the cumulative depth of bradycardia events between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Compare the cumulative duration of bradycardia events. | 24 hours
  To compare the cumulative duration of bradycardia events between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.
Nursing assessment scores -NPASS scoring system (6). | 24 hours
  To compare NPASS scores (6) between periods of presence and absence of tactile vibratory device stimulation adjunct to standard of care.

OTHER OUTCOMES:
Post trial feedback | up to 24 weeks
  To conduct post-trial surveys to gather feedback from bedside nurses and parents/legal guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Oana Dr Anton, MBBS MRCPCH, Principal Investigator — Brighton and Sussex University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Publication and conference presentation of results planned

REFERENCES:
- [Background] Kesavan K, Frank P, Cordero DM, Benharash P, Harper RM. Neuromodulation of Limb Proprioceptive Afferents Decreases Apnea of Prematurity and Accompanying Intermittent Hypoxia and Bradycardia. PLoS One. 2016 Jun 15;11(6):e0157349. doi: 10.1371/journal.pone.0157349. eCollection 2016. PMID 27304988
- [Background] Martin RJ, Di Fiore JM, Macfarlane PM, Wilson CG. Physiologic basis for intermittent hypoxic episodes in preterm infants. Adv Exp Med Biol. 2012;758:351-8. doi: 10.1007/978-94-007-4584-1_47. PMID 23080182
- [Background] te Pas AB, Davis PG, Kamlin CO, Dawson J, O'Donnell CP, Morley CJ. Spontaneous breathing patterns of very preterm infants treated with continuous positive airway pressure at birth. Pediatr Res. 2008 Sep;64(3):281-5. doi: 10.1203/PDR.0b013e31817d9c35. PMID 18458652
- [Background] Robertson CM, Watt MJ, Dinu IA. Outcomes for the extremely premature infant: what is new? And where are we going? Pediatr Neurol. 2009 Mar;40(3):189-96. doi: 10.1016/j.pediatrneurol.2008.09.017. PMID 19218032
- [Background] Henderson-Smart DJ, Steer PA. Caffeine versus theophylline for apnea in preterm infants. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000273. doi: 10.1002/14651858.CD000273.pub2. PMID 20091506
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830
- [Background] Randerath W, Verbraecken J, Andreas S, Arzt M, Bloch KE, Brack T, Buyse B, De Backer W, Eckert DJ, Grote L, Hagmeyer L, Hedner J, Jennum P, La Rovere MT, Miltz C, McNicholas WT, Montserrat J, Naughton M, Pepin JL, Pevernagie D, Sanner B, Testelmans D, Tonia T, Vrijsen B, Wijkstra P, Levy P. Definition, discrimination, diagnosis and treatment of central breathing disturbances during sleep. Eur Respir J. 2017 Jan 18;49(1):1600959. doi: 10.1183/13993003.00959-2016. Print 2017 Jan. PMID 27920092
- [Background] Shevtsova NA, Marchenko V, Bezdudnaya T. Modulation of Respiratory System by Limb Muscle Afferents in Intact and Injured Spinal Cord. Front Neurosci. 2019 Mar 26;13:289. doi: 10.3389/fnins.2019.00289. eCollection 2019. PMID 30971888
- [Background] Potts JT, Rybak IA, Paton JF. Respiratory rhythm entrainment by somatic afferent stimulation. J Neurosci. 2005 Feb 23;25(8):1965-78. doi: 10.1523/JNEUROSCI.3881-04.2005. PMID 15728836
- [Background] Dekker J, Martherus T, Cramer SJE, van Zanten HA, Hooper SB, Te Pas AB. Tactile Stimulation to Stimulate Spontaneous Breathing during Stabilization of Preterm Infants at Birth: A Retrospective Analysis. Front Pediatr. 2017 Apr 3;5:61. doi: 10.3389/fped.2017.00061. eCollection 2017. PMID 28421171
- [Background] Solkoff N, Matuszak D. Tactile stimulation and behavioral development among low-birthweight infants. Child Psychiatry Hum Dev. 1975 Fall;6(1):33-7. doi: 10.1007/BF01434430. PMID 1238237
- [Background] Lovell JR, Eisenfeld L, Rosow E, Adam J, Lapin C, Bronzino JD. Vibrotactile stimulation for treatment of neonatal apnea: a preliminary study. Conn Med. 1999 Jun;63(6):323-5. No abstract available. PMID 10432764
- [Background] Pichardo R, Adam JS, Rosow E, Bronzino J, Eisenfeld L. Vibrotactile stimulation system to treat apnea of prematurity. Biomed Instrum Technol. 2003 Jan-Feb;37(1):34-40. doi: 10.2345/0899-8205(2003)37[34:VSSTTA]2.0.CO;2. PMID 12613292
- [Background] Pietravalle A, Cavallin F, Opocher A, Madella S, Cavicchiolo ME, Pizzol D, Putoto G, Trevisanuto D. Neonatal tactile stimulation at birth in a low-resource setting. BMC Pediatr. 2018 Sep 20;18(1):306. doi: 10.1186/s12887-018-1279-4. PMID 30236090
- [Background] Frank UA, Bordiuk JM, Borromeo-McGrail V, Saltzman MB, Keitel HG. Treatment of apnea in neonates with an automated monitor-actuated apnea arrestor. Pediatrics. 1973 May;51(5):878-83. No abstract available. PMID 4703399
- [Background] Cramer SJE, Dekker J, Dankelman J, Pauws SC, Hooper SB, Te Pas AB. Effect of Tactile Stimulation on Termination and Prevention of Apnea of Prematurity: A Systematic Review. Front Pediatr. 2018 Mar 2;6:45. doi: 10.3389/fped.2018.00045. eCollection 2018. PMID 29552548
- See also: Sponsor website — http://www.inspiration-healthcare.com